CLINICAL TRIAL: NCT03848767
Title: An Early Feasibility Study to Evaluate the Functionality and Safety of an Automated Insulin Delivery System in Adult Patients With Type 1 Diabetes Mellitus During Meal Challenges
Brief Title: A Study of an Automated Insulin Delivery System in Adult Participants With Type 1 Diabetes Mellitus During Meal Challenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17177; F3Z-MC-IORD (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AID System Containing Insulin Lispro (Experimental): The AID system is comprised of a continuous subcutaneous insulin infusion (CSII) pump component with a hybrid closed-loop control (HCLC) algorithm, and a continuous glucose monitor (CGM) component.
  Interventions: Device: AID System; Drug: Insulin Lispro

INTERVENTIONS:
Device: AID System — AID System
  Other Names: LY8888AU
Drug: Insulin Lispro — Individualized doses of insulin lispro administered via the AID system to maintain glycemic control except during meal challenges.
  Other Names: LY275585

SUMMARY:
The Automated Insulin Delivery (AID) System is an investigational insulin delivery device being developed for use for participants with diabetes. The purpose of this study is to assess the safety of the AID system during meal challenges.

ELIGIBILITY:
Inclusion Criteria:

* Participants with T1DM for at least 2 years and who have used an insulin delivery system with any rapid-acting insulin analog for the preceding 6 months
* Have a body mass index of 18.5 to 37 kilogram per meter squared
* Have a hemoglobin A1c level ≥6.0% and ≤9.0%

Exclusion Criteria:

* Have known allergies or history of hypersensitivity to insulin lispro
* Have had an episode of severe hypoglycemia within the past 6 months
* Have had more than 1 episode of diabetic ketoacidosis in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | In-Patient Period (3 Days)
  Number of AEs
Continuous Glucose Monitor (CGM) Measured Percentage of Time <70 mg/dL | In-Patient Period (3 Days)
  CGM measured percentage of time <70 milligrams per deciliter (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Rainier Clinical Research Center, Renton, Washington, United States

IPD SHARING:
Plan to Share IPD: No